CLINICAL TRIAL: NCT03725150
Title: Iron Deficiency Anaemia in Pregnancy: an Observational Study of Tolerability, Compliance With Oral Iron Therapy and Effects on Haematological/Biochemical Markers
Brief Title: Treatment of Iron Deficiency Anaemia in Pregnancy Study
Acronym: TIAP
Status: Completed | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018OBS100
Record Dates: First submitted 2018-10-29; First posted 2018-10-30 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Anemia, Iron Deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The burden of anaemia remains unacceptably high during pregnancy. Over a third of women are anaemic by their third trimester of pregnancy. The most common cause is iron deficiency. One key factor is rising iron requirements throughout pregnancy. There are risks associated with anaemia for the mother and infant. Anaemia in the first and second trimester has been significantly correlated with low birth weight and pre-term birth, and is associated with impaired neurological development of the baby. It also increases the risk of intrauterine fetal death, and the likelihood of the mother requiring blood transfusions during or after delivery.This study is a prospective cohort study, which aims to better define the natural history and understand how to use oral iron therapy for iron deficiency anaemia in pregnant women. This includes documenting the impact of treatment on anaemia symptoms, side effects, and the level of success of iron therapy using several haematological tests. Pregnant women will be invited to participate in this study and treated using a treatment schedule as described in national guidelines. Additional blood samples will be taken for subsequent detailed analysis of pathways of iron metabolism to better predict the response to oral iron therapy during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (any stage during pregnancy up to 36 weeks) and women in the puerperium (within 6 weeks postdelivery) with anaemia as defined by World Health Organization (WHO) criteria and described in British Society Haematology (BSH)/ British Committee for standards in Haematology (BCSH) guidelines.

  1. First trimester < 110g/l
  2. Second and third trimester < 105g/l
  3. Puerperium < 100g/l
* Age: 18-45 years
* Agreement to participate in the study with consenting

Exclusion Criteria:

* Anaemic women presenting at or after 36 weeks as there may be insufficient time to delivery to assess responses to oral iron)
* Anaemic women affected by a (major) haemoglobinopathy e.g. B thalassaemia major sickle cell disease
* Women with overt clinical signs of sepsis
* Allergies to iron
* Hyperemesis Gravidarum / persistent vomiting
* Women with inflammatory conditions such as Crohns, ulcerative colitis, Systemic lupus erythematosus, Rheumatoid arthritis.
* Women with chronic renal failure

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Anaemic (iron-deficient) pregnant women.
Study Population: Anaemic (iron-deficient) pregnant women receiving oral iron replacement therapy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
An increase in haemoglobin of at least 10g/L | 2 to 4 weeks after the onset of iron therapy.

CONTACTS AND LOCATIONS:
Overall Officials: David Churchill, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- New Cross Hospital, Wolverhampton, West Midlands, United Kingdom